CLINICAL TRIAL: NCT04614116
Title: Cold Induced Futile Cycles In White Adipose Tissue: Quantification And Characterization With Dual Glucose Analysis
Brief Title: Cold Induced Futile Cycles In White Adipose Tissue
Acronym: Metabol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Baden (Other)
Responsible Party: Principal Investigator, Irene A. Burger, Head of clinic, Kantonsspital Baden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Cold exposure of WAT
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Metabolism Disorder
Keywords: Glucose metablism; futil cycles; FDG PET/CT
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Non blinded, randomised, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biopsy without cold induction (Other): Participants will undergo a fat biopsy after the first scan, without cooling
  Interventions: Diagnostic Test: FDG PET/CT; Diagnostic Test: 13C-Glucose injection
- Biopsy with cold induction (Other): Participants will undergo a fat biopsy after the second scan, with cooling
  Interventions: Other: External cooling; Diagnostic Test: FDG PET/CT; Diagnostic Test: 13C-Glucose injection

INTERVENTIONS:
Other: External cooling — water-circulating cooling/warming sleeves connected to a medical cooling device (Hilotherm Clinic®, Hilotherm GmbH, Germany) will be placed around the subject's abdomen and lower back. Initially the temperature of the water will be set to 25°C. A mild cold stimulus will be applied by reducing the temperature of the circulating water by approximately 1°C every 2 minutes to a minimum of 10°C.
  Arms: Biopsy with cold induction
Diagnostic Test: FDG PET/CT — o 75 MBq 18F-FDG will be injected through the intravenous line on the scanner manually (bolus injection) with a simultaneous start of dynamic FDG-PET/CT scan for 45 minutes and a partial body scan from head to the abdomen after 45 minutes. Total scan time 60 minutes.
Diagnostic Test: 13C-Glucose injection — 0.5 g 13C-Glucose i.v. infusion over 5 minutes, after termination of FDG injection

SUMMARY:
Investigation of futile cycles in white adipose tissue under cold conditions for thermogenesis using two substitutes for glucose metabolism (18F-FDG and 13C-Glucose).

DETAILED DESCRIPTION:
Thermogenesis is defined as a process, which generates heat by the depletion of energy-rich molecules. Evolutionary, it is an essential process that allows the survival at lower temperatures. Since the discovery of brown adipose tissue (BAT) it is believed that this part of the adipose tissue can dissipate energy for heat thanks to the uncoupling protein 1 (UCP1). Since energy expenditure is increased as a consequence of thermogenesis, pharmacological induction of this pathway presents an interesting therapeutic target to counter obesity. However, recent investigations indicate that white adipose tissue (WAT) is much more versatile and probably essentially indispensable for thermogenesis.

To investigate the mechanism of this futile cycle in WAT we plan to investigate the glucose metabolism in 24 healthy volunteers with 2 exams (one with and one without external cooling) with two substitutes for glucose. We will use 18F-FDG to quantify the glucose influx into WAT using dynamic PET/CT scans and 13C-Glucose to analyze the downstream metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Healthy participants, as determined by screening assessments and Principal Investigator's judgment
* Health status is defined by the absence of evidence of any active or chronic disease following a medical and surgical history, basic physical examination and blood test

Exclusion Criteria:

* any clinically relevant history or the presence of e.g. respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurological, cardiovascular, psychiatric, metabolic disease, etc.
* Intake of the following medications: Insulin, oral antidiabetic drugs, GLP-1-agonists, Corticosteroids, Sympathomimetic and Sympatholytic drug, Beta-Blocker, Statins.
* BMI > 35 kg/m2
* Resting pulse rate > 70 bpm, resting blood pressure > 130/90 mmHg.
* Serum creatinine > 145 µmol/L
* ASAT> 75 U/L and ALAT > 75 U/L
* γ GT > 100 UI/L and total bilirubin > 30 µmol/l
* Glucose > 7.1 mmol/L
* HbA1c > 46 mmol/mol (>6.4%)
* Intake of anticoagulants or inhibitors of platelet aggregation (e.g. Aspirin, clopidogrel).
* Known tendency to form keloids (hypertrophic scar tissue)
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Participation in another study involving ionizing radiation in the same year
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male volunteers
Enrollment: 24 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Comparison of FDG influx into WAT | 2 days
  Comparing the 18F-FDG influx rate (Ki) into the white adipose tissue with and without cold stimulation (intra-individually).

SECONDARY OUTCOMES:
Quantification of 13C-Glucose metabolites in fat | 2 days
  Comparing the 13C-Glucose accumulation in white adipose tissue between Group A (without cold) and B (with cold) stimulation
Quantification of 13C-Glucose metabolites in blood | 2 days
  13C-Lactate concentration in blood samples between Group A (without cold) and B (with cold) stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Irene A. Burger, MD, Principal Investigator — Kantonsspital Baden
Locations (1):
- Kantonsspitla Baden, Baden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No